CLINICAL TRIAL: NCT00640289
Title: Clinical Research Study of Factor XIII Concentrate From Human Plasma Fibrogammin P in Patients With Factor XIII Deficiency
Brief Title: Clinical Trial of Factor XIII (FXIII) Concentrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB-IND5986
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2008-03

CONDITIONS: Hemophilia; Factor XIII Deficiency
Keywords: Factor XIII Deficiency; Rare Bleeding Disorder; Hemophilia; Fibrogammin P
MeSH Terms: conditions — Hemophilia A; Factor XIII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Treatment
  Interventions: Drug: Fibrogammin P

INTERVENTIONS:
Drug: Fibrogammin P — Prophylaxis treatment

SUMMARY:
Congenital deficiency of Factor XIII is a rare but potentially life threatening disorder. It is inherited in an autosomal recessive fashion. Infusion of Factor XIII has proved to be useful for prevention and treatment of bleeding episodes, especially of spontaneous intracranial bleedings. In this study, Fibrogammin P will be given to patients with congenital Factor XIII deficiency and congenital/acquired FXIII deficiency to prevent bleeding and to treat established bleeding episodes. For Factor XIII prophylaxis to prevent hemorrhages, the dosage will depend on the weight of the subject. The frequency of Factor XIII administration will be determined by the factor's circulating half-life. During the first month only, a Factor XIII pharmacokinetic study will be determined over a 4-week period. Safety data will include accrual of information on viral safety, liver function, complete blood counts and adverse events. Historical data concerning spontaneous bleeds will be collected whenever possible two years prior to treatment with Fibrogammin P.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be of either sex or age. Children and newborn infants are specifically included in this study.
* Patient must have documented congenital Factor XIII deficiency
* Patient or legal guardian must sign informed consent
* Patients who have negative serology for hepatitis B should receive Hepatitis B vaccination.

Exclusion Criteria:

* Patient has acquired Factor XIII deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2000-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane J. Nugent, MD, Principal Investigator — Children's Hospital of Orange Co.
Locations (1):
- Children's Hospital of Orange Co., Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Factor XIII: Prophylactic dose of Factor XIII Concentrate (Human) was to be 10 to 20 U/kg b.w. administered IV over 5 minutes once every 4 weeks, and later tailored to subjects PK profile.
Period: Overall Study
Arm/Group | Factor XIII
Started | 72
Completed | 59
Not Completed | 13
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Data collected under different amendment | 2
Not completed — Transferred to another center | 1
Not completed — Missing status | 5

BASELINE CHARACTERISTICS:
Population: Safety Population (SP): The safety population consists of all subjects who received a dose of FXIII during the study. Age is age at time of first dose.
Arm/Group | Factor XIII
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (14.09)
Age, Customized [Count of Participants; unit: Participants]
  <2 years | 9
  2 to<16 years | 34
  16 to<65 years | 28
  ≥65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 48
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment of Bleeding Events Requiring Additional Factor XIII Infusions
Description: Response is defined as: Excellent/Good = adequate hemostasis, similar to that expected for subjects without known bleeding disorders; Fair/Poor = hemostasis less than expected; None = severe bleeding, judged due to disease despite Factor XIII (FXIII) therapy. Only the subjects who needed additional FXIII infusions (apart from the prophylactic treatment) to control a bleed and who had investigator assessment of efficacy were counted in this outcome.
Time Frame: Within 12 hours of FXIII infusion
Population: Safety Population (SP): The safety population consists of all subjects who received a dose of FXIII during the study.
Measure: Count of Units; unit: Number of bleeds
Units Other Than Participants: Number of bleeds
Arm/Group | Factor XIII
Number analyzed (Participants) | 22
Number analyzed (Number of bleeds) | 34
Number of bleeds
  Excellent/Good | 30
  Fair/Poor | 1
  None | 0
  Missing | 3

2. Secondary Outcome: Surgical Efficacy Assessments With Factor XIII
Description: Surgical efficacy is defined as: Excellent/Good = adequate hemostasis, similar to that expected for subjects without known bleeding disorders; Fair/Poor = hemostasis less than expected; None = severe bleeding, judged due to disease despite Factor XIII (FXIII) therapy. Only the subjects who underwent a surgical procedure were counted in this outcome measure.
Time Frame: During surgical procedure
Population: SP
Measure: Count of Units; unit: Surgical procedures
Units Other Than Participants: Surgical procedures
Arm/Group | Factor XIII
Number analyzed (Participants) | 15
Number analyzed (Surgical procedures) | 16
Surgical procedures
  Excellent/Good | 15
  Fair/Poor | 0
  None | 0
  Missing | 1

ADVERSE EVENTS:
Time Frame: 9 years
Arm/Group | Factor XIII
All-Cause Mortality (participants affected / at risk) | 3/72
Serious Adverse Events (participants affected / at risk) | 8/72
Other Adverse Events (participants affected / at risk) | 32/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Factor XIII (N=72)
Catheter related infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Gunshot wound (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Brain mass (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Suicidal behavior (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Factor XIII (N=72)
Contusion (Injury, poisoning and procedural complications) | 13 (32)
Joint injury (Injury, poisoning and procedural complications) | 7 (9)
Limb injury (Injury, poisoning and procedural complications) | 4 (10)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (22)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No